CLINICAL TRIAL: NCT02953249
Title: Wound Healing After Tooth Extraction in Individuals With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marina Helena Cury Gallottini, Professor, University of Sao Paulo
Other Study IDs: 51979315.7.0000.0075
Record Dates: First submitted 2016-03-21; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: None Retained — stimulated saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: The study group will include 30 subjects with type 1 diabetes mellitus who require extraction of 1 or more erupted teeth
- Control group: The control group will include 30 healthy subjects, without diabetes mellitus, in need of tooth extraction

SUMMARY:
Dental treatment to individuals with diabetes mellitus, particularly type 1 diabetes (T1DM), has always represented a challenge to the dentist. The literature provides some scientific evidence showing that diabetes is a risk factor for the occurrence of oral opportunistic infections, abnormal bone metabolism and delay in tissue repair, but with varying degrees of evidence.

Hyperglycemia, as well as diabetes, are known as risk factor for post-surgical infections, so maintaining the glycemic control in the postoperative period has been standard to health care. However, there are few studies on the impact of the glycemic control in the repair process after tooth extractions. And, to our knowledge, there aren't evidences that infections resulting from oral surgery are more frequent in individuals with diabetes or that the antibiotics prophylaxis is needed for these individuals before invasive dental procedures.

Some prospective studies show that people with diabetes, especially type 2 (T2DM), do not exhibit higher frequency of complications in repair process after tooth extractions compared to healthy individuals without diabetes. Recently, the study conduct by Fernandes et al., 2015, found higher frequency of delay on epithelial covering of the alveolus after 21 days of tooth extraction in individuals with T2DM, comparing to a control group. Delay was not related to infection and on the day 60th after surgery, all alveolus were totally epithelized. One of the author's hypothesis for the delay in the alveolar epithelialization on the participants with T2DM was the possible reduction of Epithelial Grow Factor (EGF) in saliva of these individuals. Some studies already demonstrated the reduction in salivary detection of EGF in individuals with diabetes.

There aren't prospective studies in the literature at our disposal, that evaluated intraoperative complications of tooth extractions of teeth already erupted in individuals with T1DM, or even post tooth extraction healing and the chronology of epithelialization of the alveolus and its relation with the degree of salivary EGF.

The aim of this study is to evaluated the intraoperative events and the post- tooth extraction healing, regarding the chronology of the repairing events and the occurrence of postoperative complications in individuals with T1DM compared to a control group. Besides, this study intend to relate the time of complete epithelial covering of the alveolus with the EGF collected by whole stimulated saliva.

DETAILED DESCRIPTION:
This prospective, longitudinal, case-control study will include 30 subjects with type 1 diabetes mellitus who require extraction of 1 or more erupted teeth, which will make part of study group (SG). Other 30 healthy subjects, without diabetes mellitus, in need of tooth extraction will make part of control group (CG). The groups will be matched by gender and age.

This project will be submitted to the Research and Ethics Committee of Dentistry College in University of Sao Paulo and all participants will sign a Consent Term.

All subjects who agreed to participate of this research will sign the Consent Term. A questionnaire will be filled by the researcher, through information obtained by direct questioning of the participant, contaning demographic data (gender, age), medical history, dental history, medications and other health problems.

After anamnesis, the researcher will make a clinical evaluation of oral health to see the necessity of tooth extractions. If there is any indication of tooth extraction, a periapical radiograph will be performed. Also, will be required complimentary blood exams with blood count, fasting glycemia and coagulation factors. Subjects that will be in use or that made use antibiotics at least a month before the tooth extraction will be excluded from this study.

On the day of the surgical procedure, will be measured, in the individuals of SG, quick exams of glicated hemoglobin (A1C) through the equipment A1C Now+ Multi-Test HbA1c System Bayer®. The glycaemia will be measured with the equipment Accu-Check®, before and after the tooth extraction and in each appointment of post-surgery (Day 3, Day 7, Day 21, Day 60). The blood pressure will also be measured before and after the tooth extraction.

The saliva collection will be performed before the surgical procedure, at least one hour after the patient has fed. It will be collected stimulated saliva through the chewing of parafilm. In the first minute the patient only will normally chew and swallow saliva, in the next five minutes all saliva produced will be deposited in a graduated Falcon tube. Salivary flow is going to be measured and expressed in mililiters per minute. The collected saliva will centrifuged at 14000 rpm for 15 minutes. The supernatant will be collected and freeze at -80oC and the sediment content will be discarded.

The saliva analysis for measuring the concentration of EGF will be carried out by immunoassay using an EGF ELISA kit (Novex®). The EGF concentration is expressed by the optical density reading of the samples compared to a standard curve, with the aid of a microplate reader with an absorption of 450nm, followed by 570nm wavelength.

The Invitrogen human EGF kit is a solid phase sandwich Enzyme Linked-Immuno-Sorbent Assay (ELISA). A polyclonal antibody specific for human EGF has been coated onto the wells of the microtiter strips provided. Samples, including standards of known human EGF content, control specimens, and unknowns, are pipetted into these wells.

During the first incubation, the Hu EGF antigen binds to the immobilized (capture) antibody on one site. After washing, a biotinylated monoclonal antibody specific for Hu EGF is added. During the second incubation, this antibody binds to the immobilized Hu EGF captured during the first incubation.

After removal of excess second antibody, Streptavidin-Peroxidase (enzyme) is added. This binds to the biotinylated antibody to complete the four-member sandwich. After a third incubation and washing to remove all the unbound enzyme, a substrate solution is added, which is acted upon by the bound enzyme to produce color. The intensity of this colored product is directly proportional to the concentration of Hu EGF present in the original specimen.

On the same day, after measuring blood pressure, glycaemia and A1C, and saliva collection, the tooth extraction will be performed. No antibiotics will be prescribed before or after surgery, as prophylactic function. Individuals of SG will be oriented to feed and administer insulin normally. Subjects with abnormal laboratorial exams or abnormal glycaemia (under 70 or above 400) will re-evaluated and the tooth extraction post-pone.

The tooth extractions will be performed by the same dentist with experience in minor oral surgery, in the Special Care dentistry center of the Dental School of University of Sao Paulo. The subjects of both groups who agreeded to participate will be submitted by conventional extraction technique, which is the same technique for any other patient of the Center. The participants will receive the same intervention of tooth extraction of patients who are not enrolled in the study, as following: after the anesthetic block will be held sindesmotomy, taking off the periodontal, tooth dislocation with the aid of lifts and removal of the tooth with forceps. The surgical technique will be modified depending on the condition of the tooth in the alveolus, performing dental section or osteotomy when necessary. Finally, curettage of the socket will be held and a simple suture with silk thread 3-0.

At the end of surgery, the blood pressure and glycaemia will be measured again. Information of the surgery procedure will be recorded, such as the tooth that was extracted, the reason of tooth was extracted (caries, periodontal disease, orthodontic needed), time spent on the surgery, number of anesthetic tubes and complications.

It will be asked for the participants to press with a gauze the alveolar region for 30 minutes to control bleeding. It will be prescript only analgesic, every 8 hours, for 3 days, in case of pain. The participant will receive postoperative written instructions.

Evaluation of repair and possible complications of the surgical wound will be held in 4 different moments, on day 3, 7, 21 and 60 after surgery. These evaluation it will always be perform by the researcher, trained and calibrated. Will be observed signs and symptoms such as edema, erythema, bone exposure, fever, pain and analgesic need. Glycaemia will be measured in all appointments from individuals from SG. Digitalized periapical radiograph will be performed at the days 7 and 60.

The repair process will be considered late when the following events do not match the period considered normal: day 3- alveolus filled by blood clot and fibrin; day 7- alveolus filled with granulation tissue; day 21- complete epithelialization of the wound; day 60- alveolus exhibiting bone deposition, radiographically observed. In case of delay in complete epithelialization after day 21, the subject will be accompanied by further consultations every 7 days for evaluation. If there is a delay in the alveolar bone deposition in the day 60, the subject will undergo another monitoring at day 90 for new radiography and evaluation.

In case of post-extraction infection (alveolitis), will set up the recommended treatment described by Kaya et al., 2011, with removal of infected debris, with abundant irrigation with saline 0.9% NaCl and curettage. It will also be prescribed antibiotics, Amoxicilin 500mg or Clindamicin 300mg, every 8 hours for 7 days, and anti-inflammatory, Nimesulide 100mg, every 12 hours for 5 days (Barasch et al., 2008).

The pain will be evaluated and assessed at the time of each appointment, through the Visual Analogue Scale (VAS), that consists of direct questioning to the patient and a visual demonstration of the scale (Annex A), being zero the total absence of pain and ten the maximum bearable level of pain by the patient.

After 60 days of surgery, the post-operative will be classified as: without complications or with complications, according to the presence or absence of signs and clinical symptoms observed. It will also be classified in: without delay and delay, according to the chronology of repair observed. According to Cheung et al., 2001, the following situations will be considered as post-operative complications:

* Acute alveolar infection: characterized by pain, erythema, edema, purulent secretion and fever;
* Acute inflammation of the alveolus: characterized by pain, inflammation, perialveolar tissue, but without purulent secretion and no fever;
* Alveolitis: characterized by persistent throbbing pain and bone exposure. All data will be transferred to an Excel spreadsheet and analyzed descriptively and associated with each other. Complications will be compared between the two groups. Additionally, in the study group, we will investigate if the occurrence of complications was related to A1C, glycaemia at surgery day, as well as EGF of saliva.

Will be held in all subjects (SG and CG) at least 3 periapical radiographs through paralleling technique, for each tooth requiring extraction. The first radiograph will be performed at the time of anamnesis, with conventional radiographic film in order to diagnose the need for extraction and assess the condition of the tooth. The second and third radiographs will be carried out using a digital sensor, at day 7 and day 60, using the digital device Soredex DIGORA Optime®, to evaluate the alveolar bone repair by grayscale concentration captured.

For standardization of these 3 X-rays of the same tooth in the same subject, a bite record of each subject will be carried out with silicone and will always be used to take the radiograph. The alveolus will be considered repaired and without delay when, at the day 60, show complete bone deposition.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 1 diabetes mellitus for study group
* Healthy individuals without diabetes mellitus for control group

Exclusion Criteria:

* under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will include 30 subjects with type 1 diabetes mellitus who require extraction of 1 or more erupted teeth
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Wound healing change after tooth extraction through epithelialization | 60 days after surgery
  Evaluation of repair and possible complications of the surgical wound will be held in 4 different moments, on day 3, 7, 21 and 60 after surgery. These evaluation it will always be perform by the researcher, trained and calibrated. Will be observed signs and symptoms such as edema, erythema, bone exposure, fever, pain and analgesic need.
  The repair process will be considered late when the following events do not match the period considered normal: day 3- alveolus filled by blood clot and fibrin; day 7- alveolus filled with granulation tissue; day 21- complete epithelialization of the wound; day 60- alveolus exhibiting bone deposition, radiographically observed.

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory values | Within 30 days before the tooth extraction
  Participants with thrombocytopenia or deficiency in coagulation factors will be re-evaluated
Adverse events that are related to the surgery | up to 3 hours before surgery
  Participants with diabetes mellitus who show moments before surgery hypoglycemia (under 100mg/dL), hyperglycemia (above 400mg/dL), hypertension or hypotension will be re-schedule.
Salivary flow | Before surgery with 5 minutes collection
  It will be calculated the salivary flow with millimeter per minute, being the study group compared to control group
Epidermal Grow Factor (EGF) | after the saliva collection of all participants the samples will be frozen at -80 Celsius degrees. The EGF of the samples will be analyzed by the end of all patients collection (after 1 years collection)
  The EGF in stimulated saliva will be analyzed and compared between groups (pg/ml)
Radiographic analysis of bone repair | Between day 7 and day 60 after tooth extraction
  Evaluate the alveolar bone repair by grayscale concentration captured using the software ImageJ

CONTACTS AND LOCATIONS:
Overall Officials: Marina HC Gallottini, Professor, Study Chair — University of Sao Paulo, Lineu prestes Ave, 2227, Sao Paulo, Brazil
Locations (1):
- Dental School of University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No